CLINICAL TRIAL: NCT05584137
Title: A Phase II Study to Evaluate the Efficacy, Safety and Tolerability of HLX26 (Anti-LAG-3 Monoclonal Antibody Injection) in Combination with Serplulimab in Patients with MCRC That Have Received 3 Prior Lines of Therapy
Brief Title: Evaluate the Efficacy, Safety and Tolerability of HLX26 and Serplulimab in Patients with MCRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor clinical trial accrual, the study was terminated.
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX26HLX10-mCRC201
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose cohort 1 of the first stage (escalation stage) (Experimental): In this cohort, HLX26 500 mg in combination with HLX10 300 mg will be intravenously administered every 3 weeks. 3 to 6 subjects will be enrolled in this cohort. Patients will be treated with investigational products until 2 years, disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first).
  Interventions:
  Drug: HLX26 Drug: HLX10
  Interventions: Drug: HLX26; Drug: HLX10
- Dose cohort 2 of the first stage (escalation stage) (Experimental): In this cohort, HLX26 800 mg in combination with HLX10 300 mg will be intravenously administered every 3 weeks. 3 to 6 subjects will be enrolled in this cohort. 3 to 6 subjects will be enrolled in this cohort. Patients will be treated with investigational products until 2 years, disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first).
  Interventions:
  Drug: HLX26 Drug: HLX10
  Interventions: Drug: HLX26; Drug: HLX10
- Dose cohort 3 of the first stage (escalation stage) (Experimental): In this cohort, HLX26 1600 mg in combination with HLX10 300 mg will be intravenously administered every 3 weeks. 3 to 6 subjects will be enrolled in this cohort. 3 to 6 subjects will be enrolled in this cohort. Patients will be treated with investigational products until 2 years, disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first).
  Interventions:
  Drug: HLX26 Drug: HLX10
  Interventions: Drug: HLX26; Drug: HLX10
- Dose cohort 1 of the second stage (expansion stage) (Experimental): In this cohort, HLX26 800 mg in combination with HLX10 300 mg will be intravenously administered every 3 weeks. 20 subjects will be enrolled in this cohort. Patients will be treated with investigational products until 2 years, disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first).
  Interventions:
  Drug: HLX26 Drug: HLX10
  Interventions: Drug: HLX26; Drug: HLX10
- Dose cohort 2 of the second stage (expansion stage) (Experimental): In this cohort, HLX26 1600 mg in combination with HLX10 300 mg will be intravenously administered every 3 weeks. 20 subjects will be enrolled in this cohort. Patients will be treated with investigational products until 2 years, disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first).
  Interventions:
  Drug: HLX26 Drug: HLX10
  Interventions: Drug: HLX26; Drug: HLX10

INTERVENTIONS:
Drug: HLX26 — Humanized Anti-Lymphocyte Activation Gene-3 Monoclonal Antibody
  Other Names: Anti-LAG-3 Monoclonal Antibody
Drug: HLX10 — Humanized Anti-Programmed Death-1 Monoclonal Antibody
  Other Names: Anti-PD-1 Humanized Monoclonal Antibody; SERPLULIMAB

SUMMARY:
This study is a phase II study to evaluate the efficacy, safety and tolerability of HLX26 and HLX10 in the treatment of patients with metastatic colorectal carcinoma that had received 3 prior therapies.

DETAILED DESCRIPTION:
This study is a phase II study to evaluate the efficacy, safety and tolerability of HLX26 and HLX10 in the treatment of patients with metastatic colorectal carcinoma that had received 3 prior therapies.

The study is composed of the first stage (escalation stage) and the second stage (expansion stage). In the first stage (escalation stage), a 3 + 3 dose escalation design will be used. Patients will receive 3 dose levels of HLX26 (500mg, 800mg, 1600mg) combined with HLX10 300mg intravenously every 3 weeks. Observation period of DLT lasts for 3 weeks after the first administration of HLX26. In the second stage, the safety and efficacy of 2 dose levels of HLX26 (800mg and 1600mg) combined with HLX10 300mg will be evaluated. Eligible subjects will be enrolled in the HLX26 800mg group and HLX26 1600mg group in sequence, 20 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed colorectal adenocarcinoma that is metastatic and unresectable.
* Has at least one measurable lesion per RECIST 1.1 as assessed by investigator.
* Has been treated with 3 prior lines of therapy for the disease and radiographically progressed on or after or could not tolerate prior therapies which include a fluoropyrimidine, oxaliplatin, irinotecan, an anti-VEGF therapy, an anti-EGFR therapy (if KRAS wild-type), regorafenib, TAS-102, fruquintinib, and BRAF inhibitor (if BRAF mutant-type).
* Submits an archival (≤ 5 years) or newly obtained tumor tissue sample that has not been previously irradiated for the determination of PD-L1 level and mismatch repair (MMR) status to meet the study requirements.
* Has an Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 to 1 within 7 days prior to first dose of study intervention.
* Has a life expectancy of at least 3 months, based on the investigator assessment.
* Has adequate organ function.

Exclusion Criteria:

* Has previously been found to have deficient MMR/microsatellite instability-high (dMMR/MSI-H) tumor status.
* The adverse reactions (except alopecia and other adverse reactions determined by the investigator to have no safety risk) of previous anti-tumor therapy have not yet recovered to ≤ grade 1 (CTCAE V5.0).
* Those who are known to have severe anaphylaxis (grade 4 or greater per CTCAE V5.0) to macromolecular protein preparations/monoclonal antibodies or to any component of the investigational product.
* Patients with any of the following unstable or poorly controlled diseases:1)Active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to the first administration of the investigational product;2)Any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (a) NYHA Class II or greater cardiac failure or left ventricular ejection fraction (LVEF) < 50%; (b) unstable angina pectoris; (c) myocardial infarction and cerebral infarction within 6 months; (d) clinically significant supraventricular or ventricular arrhythmia that has not been intervened or is poorly controlled after clinical intervention; 3)Other chronic diseases which, in the opinion of the investigator, may compromise the safety of the patient or the integrity of the study.
* Assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced.
* Previous grade 2 or greater immune pneumonia in immunotherapy; previous grade 3 or greater irAEs in immunotherapy.
* Has had other malignant tumors within 5 years before enrollment, except: (a) those with cured cervical carcinoma in situ or non-melanoma skin cancer; (b) those with cured second primary cancer without recurrence within 5 years; (c) those with double primary cancers believed to be able to benefit from this study; (d) those whose metastasis has been clearly excluded from a certain primary tumor source.
* History of prior treatment with anti-PD-1/L1, anti-CTLA-4, anti-Lag-3 antibodies or any agent targeting T cells.
* Has active autoimmune diseases (including but not limited to the following diseases or syndromes, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism), except: vitiligo or cured childhood asthma/allergy that does not need any intervention in adulthood, autoimmune mediated hypothyroidism treated with stable dose of thyroid replacement hormone, and type I diabetes treated with stable dose of insulin; those in a stable condition and requiring no systemic immunosuppressant therapy (including corticosteroid hormone) are allowed to be enrolled.
* Has received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 14 days before the first administration; Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; those with short term use of corticosteroids for prophylaxis, such as contrast agents.
* Patients in pregnancy [confirmed by serum beta-human chorionic gonadotropin (ß-HCG) test] or breastfeeding.
* Has a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or a history of organ transplantation.
* Patients with active HBV or HCV infection (HBV DNA ≥ 10*4 copies/mL or positive HCV RNA, but patients with HBV DNA < 10*4 copies / mL after treatment can be included); Subjects with co-infection of hepatitis B and hepatitis C (HBsAg or HBcAb positive, and HCV antibody positive).
* Has received live vaccines within 28 days prior to the first administration.
* Patients whose medical history or any other evidence suggests that participation in the study may confuse the results, or subjects for whom the investigator believes the study is not in their best interest.
* Participating in other clinical studies or less than 28 days from the end of the treatment of the previous clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) (the first stage) | from day1 to day 21
  The DLT of HLX26 in combination with HLX10 within 3 weeks after the first administration in patients with metastatic colorectal carcinoma.
Maximum Tolerated Dose (MTD) (the first stage) | from day1 to day 21
  The MTD of HLX26 in combination with HLX10 within 3 weeks after the first administration in patients with metastatic colorectal carcinoma.
Objective Response Rate (ORR) per RECIST 1.1 as Assessed by Investigator (the second stage) | approximately up to 6 months
  The ORR is defined as the percentage of participants who achieve a confirmed complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Overall Survival (OS) | approximately up to 24 months
  OS is defined as the time from first dose to death due to any cause.
Progression-Free Survival (PFS) per RECIST 1.1 assessed by Investigator | approximately up to 24 months
  PFS is defined as the time from first dose to the first documented disease progression per RECIST 1.1 by investigator or death due to any cause, whichever occurs first.
Duration of Response (DOR) per RECIST 1.1 assessed by Investigator | approximately up to 6 months
  DOR is defined as the time from the first documented CR or PR until disease progression or death due to any cause, whichever occurs first. DOR is only for participants who demonstrate confirmed ORR.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No